CLINICAL TRIAL: NCT04934800
Title: Oral CLADribine in Patients That Change From First-line Disease Modifying Treatments for Multiple Sclerosis: a pROspective effectivenesS and Safety Study (CLAD CROSS)
Brief Title: Prospective Effectiveness and Safety Study of Cladribine in Participants Who Change First-line DMD Treatments for Multiple Sclerosis (CLAD CROSS)
Status: Completed | Type: Observational
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Hellas sa., Greece, an affiliate of Merck KGaA, Darmstadt, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: MS700568_0070
Record Dates: First submitted 2021-06-17; First posted 2021-06-22 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cladribine; MAVENCLAD ®
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cladribine
  Interventions: Drug: Cladribine

INTERVENTIONS:
Drug: Cladribine — No intervention will be administered as a part of this study. Participants who had switched from first-line DMD treatments to treatment with cladribine tablets in routine clinical practice will be assessed for 2 years in this study.
  Other Names: MAVENCLAD ®

SUMMARY:
The main aim was to study in the real world setting the effectiveness of Cladribine tablets in terms of Annualized Relapse Rate (ARR) and disability progression, in participants who switched from a first line Disease Modifying Drug (DMD) (Interferons, Glatiramer Acetate, Teriflunomide, (Dymethyl fumarate) [DMF]) to treatment with Cladribine tablets in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with confirmed diagnosis of RRMS diagnosed by the treating physician according to applicable clinical practice guidelines -(currently McDonald 2017 criteria), with high disease activity
* Participants should have been treated with the same first-line DMD (Interferons, Glatiramer Acetate, Teriflunomide, DMF) and at a stable dose for at least one year prior to switch to Cladribine tablets and should have been prescribed Cladribine tablets, according to the decision of the treating physician, prior to enrollment in the study. Any washout period and/or washout methods required before switching (such as elimination of Teriflunomide) must have been conducted, according to the decision of the treating physician
* Required history data should be available: Multiple Sclerosis (MS) data for the 12-months pre-baseline period (annualized relapse rate); MS Medication History (prior DMDs)
* Fulfilment of the criteria for treatment with Cladribine tablets per standard of care in accordance with the local Summary of Product Characteristics (SmPC)

Exclusion Criteria:

* Contraindications to use of cladribine tablets according to the SmPC
* Participants with history of alcohol or drug abuse that could potentially interfere with their participation in the study
* Participants that have received Cladribine in the past
* Concurrent participation in an investigational study in which participant assessment and/or treatment may be dictated by a protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a confirmed diagnosis of Highly Active Relapsing-Remitting Multiple Sclerosis (RRMS).
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (61):
- Austria (3):
  - KH der Barmherzige Brüder Eisenstadt - Neurology, Eisenstadt
  - Dr. Reinhard Krendl-Head, Sankt Veit an der Glan
  - Klinik Florisdorf, Vienna
- Greece (18):
  - University of Thrace, Medical School - Neurology Department, Alexandroupoli
  - 251 General Air Force Hospital, Athens
  - 417 NIMITS Hospital, Athens
  - Aeginiteion Hospital, University of Athens - A' Neurology Department, Athens
  - Attikon University Hospital, Athens
  - Evangelismos Hospital - Neurology Department, Athens
  - Genaral Hospital of Elefsina "Thriasio", Athens
  - General Hospital of Athens "Evangelismos", Athens
  - University of Ioannina - Neurology Department, Ioannina, Ioannina
  - University General Hospital of Larissa - Rheumatology Clinic, Larissa
  - Iatriko Palaioy Faliroy, Medical Center - Neurology Department, Palaió Fáliro
  - General Hospital of Patra "Agios Andreas", Pátrai
  - University General Hospital of Patra, Pátrai
  - AHEPA General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
  - Interbalkan Hospital of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital Thessaloniki, Thessaloniki
  - St Luke's Hospital, Thessaloniki
- Italy (19):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII) - Dipartimento di Neurologia, Bergamo
  - Fondazione Istituto G.Giglio di Cefalù - Neurologia-Centro Sclerosi Multipla, Cefalù
  - Università degli Studi G. D'Annunzio, Chieti
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna - Neurologia, Cona
  - Ospedali Riuniti di Foggia - Neurology, Foggia
  - Azienda Socio Sanitaria Territoriale della Valle Olona (presidio di Gallarate) - Neurologia 2 - Sclerosi Multipla, Gallarate
  - Ospedale San Luca - S.C.Oncologia, Lucca
  - ASL 1 Avezzano L'Aquila Sulmona- Ospedale Regionale San Salvatore - Dipartimento di Neurologia, L’Aquila
  - IRCCS Centro Neurolesi Bonino Pulejo - U.O. di Neurofisipatologia ed Ambulatori, Messina
  - Azienda Ospedaliera di Rilievo Nazionale A. Cardarelli - U.O.S. Malattie Degenerative del S.N.C., Napoli
  - Ospedale Maggiore della carità - Novara, Novara
  - Centro di Riferimento Regionale per la Sclerosi Multipla (CRESM) - SCDO Neurologia, Orbassano
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone - Dipartimento di Neuroscienze, Palermo
  - Azienda Ospedaliera di Udine Ospedale S. Maria della Misericordia - UO Neurologia, Perugia
  - Grande Ospedale Metropolitano "Bianchi Melacrino Morelli - Centro Regionale Epilessia, Reggio Calabria
  - Azienda Ospedaliera San Filippo Neri - Neurologia, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza - Dip. di Neurologia e Psichiatria (servizio EMG), Roma
  - A. O. U. San Giovanni Di Dio e Ruggi D'Aragona - Struttura Complessa di Oculistica, Salerno
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma) - D.U.Neurologia, Verona
- Norway (3):
  - Vestre Viken HF Drammen Sykehus - former Sykehuset Buskerud, Drammen
  - Sykehuset Namsos, Namsos
  - Oslo Universitetssykehus HF - Ullevål, Oslo
- Poland (7):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku - Dept of Neurology, Bialystok
  - Szpital Specjalistyczny im. L.Rydygiera w Krakowie - Neurology Department, Krakow
  - Szpital Uniwersytecki w Krakowie - Uniwersytet Jagiellonski Collegium Medicum, Krakow
  - Szpital Kliniczny im.Heliodora Swiecickiego Uniwersytetu Medycznego im.K. Marcinkowskiego w Poznaniu - Dept of Neurology, Poznan
  - Pomorski Uniwersytet Medyczny - Klinika Neurologii, Szczecin
  - Wojskowy Instytut Medyczny - Klinika Neurologiczna, Warsaw
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 3 w Rybniku, Żory
- Portugal (6):
  - Centro Hospitalar de Lisboa Ocidental, E.P.E. - Hospital de Egas Moniz - Serviço de Neurologia, Lisbon
  - Unidade Local de Saúde de Matosinhos, EPE (Hospital Pedro Hispano) - Serviço de Neurologia, Matosinhos Municipality
  - Centro Hospitalar de São João, E.P.E. - Serviço de Neurologia, Porto
  - Hospital Garcia de Orta, EPE - Serviço de Neurologia, Pragal
  - Centro Hospitalar de Setubal, EPE - Hospital São Bernardo, Setúbal
  - Unidade Local de Saúde do Alto Minho, EPE - Serviço de Neurologia, Viana de Castelo
- Switzerland (5):
  - Inselspital - Universitaetsspital Bern - Neuropsychologische Rehabilitation, Neurologie, Bern
  - (CHUV), Centre Hospitalier Universitaire Vaudois - Departement des Neurosciences Cliniques, Lausanne
  - Luzerner Kantonsspital - Zentrum fuer Neurologie und Neurorehabilitation, Lucerne
  - Ospedale Regionale di Lugano - Neurologia, Lugano
  - Hôpital Régional Sion-Hérens-Conthey - Neurologie, Sion

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0070
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cladribine: Participants with relapsing-remitting multiple sclerosis who had switched from first-line disease-modifying drug (DMD) treatments to cladribine tablets as part of routine clinical practice. No intervention was administered as part of this study.
Period: Overall Study
Arm/Group | Cladribine
Started | 256
Completed | 234
Not Completed | 22
Not completed — Other | 1
Not completed — Withdrawal by Subject | 5
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 9
Not completed — Lost to Follow-up | 5
Not completed — Enrolled but not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cladribine
Number analyzed (Participants) | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174
  Male | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 256
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 253
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Annualized Relapse Rate (ARR) Between the Pre-Baseline 12-Month Period (Baseline) and Over the 12 Months Period Before the End of Study Follow-Up (2 Years)
Description: ARR defined as the number of relapses per year. A relapse was defined as the appearance of new symptoms or the exacerbation of pre-existing symptoms that were attributed to Multiple Sclerosis (MS) and occurred over a minimum of 24 hours and separated from a previous attack by at least 30 days, in the absence of fever or infection. Baseline ARR was defined as the total number of relapses reported in the last 12 months prior to Cladribine treatment. ARR 12-months prior to End Of Study was calculated as the sum of the number of MS relapses reported at Visit 3 and Visit 4 divided by the number of days between Visit 4 date and Visit 2 date and multiplied by 365.25. For a change from baseline, 95 percent (%) Confidence Interval (CI) for the difference were presented together with summary statistics. These CIs were included as a descriptive measure of effect.
Time Frame: 12-months pre-baseline (Baseline) and 12 Months Prior to End of Study follow up (2 years)
Population: The Full Analysis Set (FAS) included all the participants who provided informed consent and who received at least one dose of Cladribine. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Cladribine
Number analyzed (Participants) | 221
relapses per year | -1.12 [-1.23 to -1.00]

2. Secondary Outcome: Change in ARR Between the Pre-Baseline 12-Month Period (Baseline) and Over the 12 Months Period After the Start of Cladribine (1 Year)
Description: ARR defined as the number of relapses per year. A relapse was defined as the appearance of new symptoms or the exacerbation of pre-existing symptoms that were attributed to MS and occurred over a minimum of 24 hours and separated from a previous attack by at least 30 days, in the absence of fever or infection. ARR 12-months after start of Cladribine was calculated as the sum of the number of MS relapses reported at Visit 1 and Visit 2 divided by the number of days between Visit 2 date and Cladribine start date and multiplied by 365.25.For a change from baseline, 95% CIs for the difference were presented together with summary statistics. These CIs were included as a descriptive measure of effect.
Time Frame: 12-month pre-baseline period (baseline) and over the 12 months period after start of Cladribine treatment (1 year)
Population: The FAS included all the participants who provided informed consent and who received at least one dose of Cladribine.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Cladribine
Number analyzed (Participants) | 256
relapses per year | -1.01 [-1.13 to -0.89]

3. Secondary Outcome: Percentage of Participants With 6-Month Disability Progression Measured With Expanded Disability Status Scale (EDSS)
Description: EDSS assessed disability in 8 functional systems. It was a scale based on a standardized EDSS neurological examination, which comprised optic, brain stem, pyramidal, cerebellar, sensory, and cerebral functions, as well as walking ability. An overall score ranged from 0 (normal) to 10 (death due to MS) was calculated. Progression on EDSS was defined as at least a 1-point increase in the score or an increase of at least 1.5 points if the baseline EDSS score was 0.
Time Frame: At EOS (24 months follow-up)
Population: The FAS included all the participants who provided informed consent and who received at least one dose of Cladribine. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 197
percentage of participants | 1.6 [0.43 to 3.95]

4. Secondary Outcome: Percentage of Participants With Overall 6-Month Disability Progression Measured With EDSS, Timed 25 Foot Walk (T25FW) or 9 Hole Peg Test (9HPT)
Description: Disability progression was assessed if at least one assessment (EDSS, T25FW or 9HPT) was available. As per definition, disability progression was derived as "Yes" if at least one of the below cases occured: 1. Visit 4 EDSS is greater than (>=) equal to (≥) 1 point >= Visit 3 EDSS if Visit 3 EDSS is > 0; 2. Visit 4 EDSS is 1.5 or > when Visit 3 EDSS is 0; 3. 20% increase in the T25FW score (average of the two trials) from Visit 3 to Visit 4; 4. 20% increase in the 9HPT score (The two trials for each hand are averaged, converted to the reciprocals of the mean times for each hand and then the two reciprocals are averaged) from Visit 3 to Visit 4. If none of those cases occurred, disability progression will be set to "No". The percentage of participants with 6-month disability progression at the EOS was presented including associated 95% Clopper Pearson exact intervals.
Time Frame: At EOS (24 months follow-up)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 198
percentage of participants | 4.7 [2.45 to 8.04]

5. Secondary Outcome: Percentage of Participants With 6-Month Disability Improvement Measured With EDSS
Description: EDSS assessed disability in 8 functional systems. It was a scale based on standardized neurological examination which comprised of optic, brain stem, pyramidal, cerebellar, sensory & cerebral functions, as well as walking ability. An overall score ranged from 0 (normal) to 10 (death due to MS) was calculated. Improvement on EDSS was defined as a decrease in EDSS by at least 1 point (1.5 points if baseline EDSS was 1.5).
Time Frame: At EOS (24 months follow-up)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 197
percentage of participants | 1.6 [0.43 to 3.95]

6. Secondary Outcome: Percentage of Participants With Overall 6-Month Disability Improvement Measured With EDSS, Timed 25 Foot Walk (T25FW) or 9 Hole Peg Test(9HPT)
Description: Disability improvement was assessed if at least one assessment (EDSS, T25FW or 9HPT) was available. As per definition, disability improvement was derived as "Yes" if at least one of the below cases occur:1. Visit 4 EDSS is ≥1 point smaller than Visit 3 EDSS if Visit 3 EDSS is greater than 1.5;2. Visit 4 EDSS is 0 when Visit 3 EDSS is 1.5;3. 20% decrease in the T25FW score (average of the two trials) from Visit 3 to Visit 4;4. 20% decrease in the 9HPT score (The two trials for each hand are averaged, converted to the reciprocals of the mean times for each hand and then the two reciprocals are averaged) from Visit 3 to Visit 4. If none of those cases occurred, disability improvement was set to "No". The percentage of participants with 6-month disability improvement at the end of study was presented including associated 95% Clopper Pearson exact intervals.
Time Frame: At EOS (24 months follow-up)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 197
percentage of participants | 4.7 [2.45 to 8.04]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, regardless if it is considered related to the medicinal product. Serious AE: AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs are defined as AEs that were reported or worsened on or after start of study drug dosing through the Safety Follow-up Visit. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: From start of study up to 2 years
Population: The FAS included all the participants who provided informed consent and who received at least one dose of Cladribine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 256
Participants
  TEAEs | 90
  TESAEs | 10

8. Secondary Outcome: Quality of Life as Assessed by Multiple Sclerosis Impact Scale (MSIS-29) Score: Physical and Psychological Impact
Description: MSIS-29 was a 29-item self-report measure with 20 items related to physical scale and 9 items with psychological scale. All items have 5 options:1-not at all to 5-extremely. Each of2 scales are scored by summing responses across items, converting to 0-100 scale where 100 indicates great impact of disease on daily function (worse health). Physical impact score computed by summing items 1-20 inclusive (observed score). This score was then transformed to a score on a scale of 0-100 using the formula:[100 multiplied by(observed score minus(-)20)] divided by(100-20). The psychological impact score was computed by summing items number21-29 inclusive(observed score). This score was then transformed to score on scale of 0-100 using the formula:[100 multiplied by(observed score minus 9)]divided by(45-9). Total score range ranges from 0-100, lower total score shows less psychological/physical-related impact while a higher total score indicated greater psychological/physical-related impact.
Time Frame: Baseline, Months 12 and 24
Population: The FAS included all the participants who provided informed consent and who received at least one dose of Cladribine. . Here "Number Analyzed" signifies those participants who were evaluable at specific timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine
Number analyzed (Participants) | 256
units on a scale
  Psychological Impact: Baseline | 30.8 (23.30)
  Psychological Impact: Month 12: number analyzed (Participants) | 182
  Psychological Impact: Month 12 | 24.8 (21.33)
  Psychological Impact: Month 24: number analyzed (Participants) | 148
  Psychological Impact: Month 24 | 23.7 (21.09)
  Physical Impact: Baseline | 20.1 (19.99)
  Physical Impact: Month 12 | 17.4 (17.09)
  Physical Impact: Month 24 | 17.2 (19.19)

9. Secondary Outcome: Quality of Life as Assessed by EuroQol Quality of Life Questionnaire 5 Dimensions 3 Levels (EQ-5D-3L)
Description: Quality of Life was measured using the EQ-5D-3L questionnaire. The EQ-5D-3L asks participants to rate the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ-5D-5L VAS was used to record a participants rating for his/her current health-related quality of life state and captured on a vertical VAS (0-100), where 0 =worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline, Months 12 and 24
Population: The FAS included all the participants who provided informed consent and who received at least one dose of Cladribine. Here "Number Analyzed" signifies those participants who were evaluated at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine
Number analyzed (Participants) | 256
units on a scale
  Baseline: number analyzed (Participants) | 254
  Baseline | 73.6 (19.07)
  Month 12: number analyzed (Participants) | 184
  Month 12 | 78.9 (15.17)
  Month 24: number analyzed (Participants) | 148
  Month 24 | 78.4 (17.17)

10. Secondary Outcome: Treatment Satisfaction as Assessed by Treatment Satisfaction Questionnaire for Medication Version 1.4 (TSQM v1.4) Scale
Description: TSQM version 1.4 was a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. It comprises of 14 items assessing the following 4 domains: effectiveness (questions: 1-3), side effects (questions: 4-8), convenience (questions: 9-11), global satisfaction (questions:12-14). Global Satisfaction- Question 12 scored as 1 (not at all confident) to 5 (extremely confident); question 13 scored as 1 (not at all certain) to 5 (extremely certain); and question 14 scored as 1 (extremely dissatisfied) to 7 (extremely satisfied). The scores of the domain were added together and an algorithm was used to create a score of 0 to 100. Higher scores indicated greater satisfaction.
Time Frame: Months 6, 12, 18 and 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cladribine
Number analyzed (Participants) | 256
units on a scale
  Global Satisfaction: Month 6: number analyzed (Participants) | 172
  Global Satisfaction: Month 6 | 71.3 (17.78)
  Global Satisfaction: Month 12: number analyzed (Participants) | 182
  Global Satisfaction: Month 12 | 75.4 (18.81)
  Global Satisfaction: Month 18: number analyzed (Participants) | 121
  Global Satisfaction: Month 18 | 75.0 (20.06)
  Global Satisfaction: Month 24: number analyzed (Participants) | 149
  Global Satisfaction: Month 24 | 77.2 (19.82)
  Effectiveness: Month 6: number analyzed (Participants) | 172
  Effectiveness: Month 6 | 71.7 (20.56)
  Effectiveness: Month 12: number analyzed (Participants) | 182
  Effectiveness: Month 12 | 72.6 (22.04)
  Effectiveness: Month 18: number analyzed (Participants) | 121
  Effectiveness: Month 18 | 72.3 (21.68)
  Effectiveness: Month 24: number analyzed (Participants) | 149
  Effectiveness: Month 24 | 77.5 (18.62)
  Side Effects: Month 6: number analyzed (Participants) | 169
  Side Effects: Month 6 | 96.6 (11.87)
  Side Effects: Month 12: number analyzed (Participants) | 178
  Side Effects: Month 12 | 96.1 (13.45)
  Side Effects: Month 18: number analyzed (Participants) | 119
  Side Effects: Month 18 | 96.8 (11.65)
  Side Effects: Month 24: number analyzed (Participants) | 143
  Side Effects: Month 24 | 97.2 (11.27)
  Convenience: Month 6: number analyzed (Participants) | 172
  Convenience: Month 6 | 84.4 (13.77)
  Convenience: Month 12: number analyzed (Participants) | 182
  Convenience: Month 12 | 87.9 (13.97)
  Convenience: Month 18: number analyzed (Participants) | 121
  Convenience: Month 18 | 86.3 (13.26)
  Convenience: Month 24: number analyzed (Participants) | 149
  Convenience: Month 24 | 88.9 (12.20)

11. Secondary Outcome: Number of Participants With Treatment Adherence
Description: According to the World Health Organization (WHO), treatment adherence is defined as both compliance (taking the medication in the correct dose and according to the schedule prescribed) and persistency (maintenance of the drug regimen over the long-term). Adherence to treatment, calculated as 100 × Taken tablets/Prescribed tablets
Time Frame: Up to Month 24
Population: The FAS included all the participants who provided informed consent and who received at least one dose of Cladribine. . Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 234
Participants
  90%-100% | 232
  Missing | 2

ADVERSE EVENTS:
Time Frame: From start of study up to 2 years
Description: Other AEs includes both serious and non-serious AEs as no separate NSAEs were calculated in the study.
Arm/Group | Cladribine
All-Cause Mortality (participants affected / at risk) | 0/256
Serious Adverse Events (participants affected / at risk) | 10/256
Other Adverse Events (participants affected / at risk) | 90/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine (N=256)
Appendicitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Multiple sclerosis relapse (Nervous system disorders) | 3
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine (N=256)
COVID-19 (Infections and infestations) | 24
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 3
Influenza (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Coronavirus infection (Infections and infestations) | 1
Dysentery (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Varicella zoster virus infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 10
Multiple sclerosis relapse (Nervous system disorders) | 9
Dizziness (Nervous system disorders) | 3
Occipital neuralgia (Nervous system disorders) | 2
Sensory disturbance (Nervous system disorders) | 2
Central nervous system lesion (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Lhermitte's sign (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 24
Leukopenia (Blood and lymphatic system disorders) | 1
Hepatic enzyme increased (Investigations) | 2
Transaminases increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
CD4 lymphocytes decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
SARS-CoV-2 test positive (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 5
Pyrexia (General disorders) | 2
Pain (General disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Depression (Psychiatric disorders) | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Deafness (Ear and labyrinth disorders) | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 1
Vision blurred (Eye disorders) | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal colic (Renal and urinary disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04934800/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT04934800/SAP_001.pdf